CLINICAL TRIAL: NCT03119220
Title: Applying a Stress Framework to Health Behavior Change: A Fitbit Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brandeis University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 15138; P30AG048785 (NIH)
Record Dates: First submitted 2017-04-13; First posted 2017-04-18 (Actual); Last update posted 2017-04-19 (Actual); Status verified 2017-04

CONDITIONS: Adult Disease
MeSH Terms: conditions — Disease

STUDY DESIGN:
Intervention Model Description: The overall behavior change goal is defined as increasing physical activity by 15% every other week over 10 weeks based on an initial one week of activity recording establishing an individual's baseline. This will result in a doubling of the initial steps by weeks 10-11, while keeping the demands and goals comparable between individuals. After the first week, informational support will be manipulated by providing one group with information in the form of physical activity monitoring only. The second group will additionally receive individualized information on how to change behavior by providing maps of a participant's neighborhood with distances depicted in steps, lists with age- and health-status appropriate suggestions as to how to increase numbers of steps, as well as medical information linking changes in physical activity to change in health outcomes; and information on health effects of behavior change by monitoring changes in sleep in conjunction with physical activity changes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low informational support (Other): After the first week, informational support will be manipulated by providing one group with information in the form of physical activity monitoring only.
  Interventions: Device: Fitbit One
- high informational support (Other): The second group will additionally receive individualized information on how to change behavior by providing maps of a participant's neighborhood with distances depicted in steps, lists with age- and health-status appropriate suggestions as to how to increase numbers of steps, as well as medical information linking changes in physical activity to change in health outcomes; and information on health effects of behavior change by monitoring changes in sleep in conjunction with physical activity changes.
  Interventions: Device: Fitbit One

INTERVENTIONS:
Device: Fitbit One — Participants will receive a Fitbit device and a detailed user manual as well as diary materials to record daily steps taken, miles walked, and flight of stairs walked for a total of 12 weeks. An in-person follow-up meeting will be scheduled 7 days after the initial meeting to establish the baseline activity level of the participant and to determine the target number of daily steps for the subsequent 5 blocks of 2 weeks.

SUMMARY:
The current study aims to counteract perceived stress-related barriers to implementation and maintenance of positive health behavior change (i.e., increasing physical activity), by providing an individually tailored and comprehensive informational support program. This translates into an intervention that, in addition to behavior monitoring (low informational support), will provide comprehensive informational support by combining advice and suggestions on how to achieve positive physical activity change with information on the health effects of such a change (high informational support). The latter will be achieved by providing information on general health benefits of increasing physical activity as well as on how physical activity change is linked to individual changes in health-relevant outcomes (i.e., mood and sleep quality changes). Specifically, it is hypothesized that:

* Higher chronic stress levels in general as well as stress perceived by the anticipated task of improving physical activity will be negatively associated with physical activity changes.
* Participants receiving informational support will show decreases in task-related stress.
* Furthermore, participants who receive comprehensive informational support will show larger physical activity improvements than participants who do not receive informational support.
* Initial stress will act as a moderator of the effects of informational support on physical activity, such that higher initial stress will reduce the positive effects of informational support.

Importantly, the proposed intervention is specifically designed to support the subsequent development of an intervention program that is not only feasible, but easy to implement by individuals motivated to achieve a positive health behavior change. A key factor will be the insights gained into stress as a mechanism that counteracts implementation and maintenance of behavior change. This is especially important given the central role of stress in negative health outcomes associated with lack of physical activity, such as poor sleep, negative mood, and chronic low-grade inflammation.

DETAILED DESCRIPTION:
Research to date has not fully addressed the role of stress in behavior change. Stress is implicated in many negative health outcomes, including poor sleep, depressive mood, and health problems related to chronic low-grade inflammation, such as hypertension, diabetes, and obesity. These negative health outcomes can lead an individual to form intentions to change health behavior. However, while stress-related negative health outcomes may motivate the attempt to change behavior, the simple intention or very attempt to change behavior may induce stress. Thus, a vicious cycle is started in which stress contributes to health conditions that necessitate and motivate behavior change attempts, while simultaneously immobilizing one from successfully implementing behavior change.

The multiple pathways through which stress can influence health behaviors may become especially apparent in middle-aged and older adults. Not only does poor health increase the urgency for behavior change and thus present a perceived threat, but the lack of resources, such as knowledge of how to implement change, and presence of barriers, such as limited time due to stressful jobs, fear of negative effects, potential to fail, or uncertainty of beneficial outcomes, all contribute to making behavior change a daunting and stressful endeavor. Conversely, many behavior change techniques can be conceptualized as stress management techniques. These techniques can operate by reducing threat perception and/or increasing access to resources, often via provision of informational support.

The proposed study thus seeks to reduce stress in order to facilitate implementation of physical activity change. This will be accomplished by providing health behavior-relevant informational support to sedentary middle-aged and older adults. Specifically, the study's aims are:

* To determine whether providing individually tailored and comprehensive informational support can increase the number of daily steps in middle-aged and older adults in a 12-week physical activity intervention setting.
* To assess how initial stress, initial stress perceived due to the intention to implement behavior change, and changes in perceived stress throughout the intervention affect physical activity change.
* To elucidate downstream effects of the intervention in terms of mental health (i.e., depressive symptoms, chronic stress) and physical health outcomes (i.e., inflammatory status) In line with the Roybal Center Aim 1, the current study explicitly targets a population of sedentary middle-aged and older adults who unsuccessfully attempted to increase physical activity. Pressure to change behavior will in many cases stem from health decrements. Furthermore, participants will be recruited from the Waltham community, which will allow targeted advertisement to ensure a diverse sample in terms of socioeconomic background as well as ethnicity. Lastly, only participants who cannot walk for stretches of several minutes without pain will be excluded, allowing individuals in early stages of disability to participate. Using a stress framework to develop the current intervention and assessing psychological, social, and biological correlates will contribute to Roybal Center Aim 2, as the findings will advance theory and empirical findings on behavior change processes and mechanism. Lastly, the current study addresses Roybal Center Aim 3, as knowledge gained from the current study will facilitate larger-scale physical activity interventions expected to improve health and quality of life of older adults.

ELIGIBILITY:
Inclusion Criteria:

* residents of Waltham and surrounding communities
* between the ages of 50 and 70+
* English and non-English speaking participants
* individuals who are sedentary and/or dealing with health issues and have been unsuccessful in implementing behavior change **We will ask participants three questions that will be rated on a 1 to 10 scale. They will be asked 1) how concerned they are about their current level of exercise, 2) how much pressure they feel to exercise more, and 3) how difficult it feels to overcome obstacles to exercise. To be eligible, participants must rate the first question at a 6 or higher and the three questions together at 15.

Exclusion Criteria:

* Participants who have been told not to participate in physical activity or who have doubts about their ability to safely increase physical activity
* not able to walk or not able to walk continuously for several minutes without pain
* being very active and rate the question regarding how much they are in motion during the day at 8 or higher (on a scale of 1-10)

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2015-05-08 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
daily steps | 12 weeks
  daily physical activity measured in steps taken

IPD SHARING:
Plan to Share IPD: Yes